CLINICAL TRIAL: NCT04718363
Title: Effects of Foam Roller Application Prior to Proprioceptive Neuromuscular Facilitation Stretching on Hamstring Flexibility and Thigh Skin Temperature in Healthy Subjects
Brief Title: Effects of Foam Rolling Prior to PNF Stretching on Hamstring Flexibility and Thigh Skin Temperature in Healthy Subjects
Acronym: PNF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sinem Yenil, Principal Investigator, PT, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4742-GOA
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: hamstring muscles; PNF stretching; foam rolling; thermal imaging; flexibility; range of motion; vibration
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PNF stretching group (Experimental)
  Interventions: Other: PNF stretching
- Non-vibration foam rolling prior to PNF stretching group (Experimental)
  Interventions: Other: Non-vibration foam rolling prior to PNF stretching
- Vibration foam rolling prior to PNF stretching group (Experimental)
  Interventions: Other: Vibration foam rolling prior to PNF stretching
- Control Group (No Intervention)

INTERVENTIONS:
Other: PNF stretching — A contract-relax PNF stretching technique will be applied to hamstring muscle.
  Arms: PNF stretching group
Other: Non-vibration foam rolling prior to PNF stretching — Prior to PNF stretching, participant will perform unilateral hamstring non-vibration foam rolling.
  Arms: Non-vibration foam rolling prior to PNF stretching group
Other: Vibration foam rolling prior to PNF stretching — Prior to PNF stretching, participant will perform unilateral hamstring vibration foam rolling (48 Hz).
  Arms: Vibration foam rolling prior to PNF stretching group

SUMMARY:
There is no study investigating the hamstring flexibility and skin temperature after combined warm-up techniques especially PNF and foam rolling. The main purpose of this study is to investigate the effects of foam roller application prior to proprioceptive neuromuscular facilitation stretching on hamstring flexibility and thigh skin temperature in healthy subjects.Secondly, it is aimed to compare the effects between non-vibration foam rolling and vibration foam rolling on measured parameters.

DETAILED DESCRIPTION:
In this study forty-eight subjects will be voluntarily recruited into the study according to inclusion criteria. Participants will be randomly assigned to Vibration Foam Rolling + PNF stretching, Non-Vibration Foam Rolling + PNF stretching, only PNF stretching and control group. Subjects will be evaluated before, immediately after and 30 minutes after intervention. Hamstring flexibility will be evaluated with Active Knee Extension Angle (AKEA) Test and functionally Sit and Reach test. Thigh skin temperature will be evaluated with thermographic imaging.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Having limitation of 20 degrees or more in knee extension angle in AKEA test,
* Right side lower extremity dominance

Exclusion Criteria:

* History of lower extremity injury in the last 12 months
* Having neurological or psychological problem
* Doing a stretching based exercise recently
* History of pain in the lower body and extremity in the Nordic Musculoskeletal Questionnaire
* Having lower extremity deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in hamstring flexibility | Change from baseline hamstring flexibility at immediately after intervention and 30 minutes after intervention
  Active Knee Extension test in supine position will be performed to measure hamstring flexibility.
Change in thigh skin temperature | Change from baseline skin temperature at immediately after intervention and 30 minutes after intervention
  Posterior thigh skin temperature will be evaluated using thermographic imaging with infrared thermal camera.
Change in functional hamstring flexibility | Change from baseline functional hamstring flexibility at immediately after intervention and 30 minutes after intervention
  Sit-and-Reach test will be performed to measure functional hamstring flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)